CLINICAL TRIAL: NCT01779804
Title: The Effect of Triage-Based Application of the Ottawa Ankle and Foot Rules (OAR/OFR) on the Number of Radiographs Ordered: A Pilot Study
Brief Title: Triage-Based Application of OFAR on the Number of Radiographs Ordered
Acronym: OFAR
Status: Completed | Type: Observational
Sponsor: Lehigh Valley Hospital (Other)
Responsible Party: Principal Investigator, Marna Rayl Greenberg, Director of Emergency Medicine Research, Lehigh Valley Hospital
Other Study IDs: PR000000185
Record Dates: First submitted 2013-01-22; First posted 2013-01-30 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2014-06

CONDITIONS: Ankle Injuries; Foot Injuries
Keywords: foot , ankle, injury
MeSH Terms: conditions — Ankle Injuries; Foot Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with foot and ankle injury: After baseline data is obtained a cohort of patients with acute foot and ankle injuries will have OFAR applied
  Interventions: Procedure: OFAR

INTERVENTIONS:
Procedure: OFAR — OFAR

SUMMARY:
Foot and ankle injuries account for nearly two million visits to Emergency Departments (EDs) in the United States and Canada each year. Of these injured patients, only 15% are diagnosed with actual fractures of the ankle. Due to such a small percentage, the "Ottawa Ankle and Foot Rules" (OFAR) were developed, which are a set of clinical decision-making guidelines that have been shown to be effective in diagnosing ankle and foot fractures. These rules are internationally accepted by the medical community, but are inconsistently applied.

At Lehigh Valley Health Network (LVHN), the ED triage nurses are routinely trained in how to use the Ottawa Ankle and Foot Rules, but the rules are not always applied which may result in unnecessary X-rays. These guidelines are current network "standard of care" (usual, established care) that allow nurses to decide treatment for foot and ankle injury patients; in other words, whether to send these patients for an X-ray or not.

The research staff is conducting this study in order to find out if using these nurse-directed guidelines--on a regular and consistent basis--can decrease the number of X-rays ordered, decrease patient waiting times/length of stay (LOS) and increase patient satisfaction with their care in the ED.

STUDY PURPOSE:

The two main goals of this study are to find out if use of the Ottawa Ankle and Foot Rules by triage nurses can decrease the amount of X-rays ordered in the ED, as well as LOS.

Secondary study goals are to: 1) see how many X-rays are ordered by physicians and physicians' assistants after patients are evaluated by the Ottawa Ankle and Foot Rules as not having had a fracture; and 2) evaluate patient and provider satisfaction with the care provided both when the Ottawa Foot and Ankle Rules are used and when they are not.

DETAILED DESCRIPTION:
Study Variables:

This study's independent variable (or "intervention/predictor" variable) is the triage application of the OAR and OFR. Dependent variables (or "outcome" variables) include the number of X-rays ordered and LOS (co-primary outcomes), and measured patient and provider satisfaction (secondary outcomes). The Principal Investigator will create and validate his own study tool/survey to measure patient and provider satisfaction.

Confounding Variables:

Confounding variables include, but are not limited to: Patient age; patient gender; census volume on the days the study is conducted; assistance from ED staff from either site; difficulty in achieving enrollment goals in a timely fashion; season of the year (i.e., skateboarding versus skiing injuries); patient expectations about their ED care; and/or patient insurance status.

Study Design/Methods:

This study is designed to be a pilot, prospective, 2-stage study to examine the application of OAR/OFR at the 17th and Chew, and Cedar Crest site EDs that aims to determine if triage nursing application of these clinical decision rules can decrease the amount of radiographs ordered, as well as decrease patient LOS.

ELIGIBILITY:
Inclusion Criteria:

* Pt must be 16 years of age (patients below 18 must be assented)
* Pt must not be pregnant
* Pt must have an isolated traumatic ankle or foot injury
* Pt must be outpatients (not admitted or assigned to observation)
* Pt must be able to speak English or Spanish
* Pt must be competent and able to give consent, (not in critical condition, intoxicated or otherwise incapacitated)
* Pt must have no neurovascular (nerve/blood vessel) compromise
* Pt must have no open fracture or visible limb deformity
* Pt must not be a pediatric patient who presents with a gait abnormality of unknown origin.

Exclusion Criteria:

* Pt must not be under the age of 16
* Pt must not be pregnant
* Pt must not have a non-isolated traumatic ankle or foot injury
* Pt must not be inpatients (may not be admitted or assigned to observation)
* Pt must not be unable to speak English or Spanish
* Pt must not be incompetent and unable to give consent, (in critical condition, intoxicated, or otherwise incapacitated)
* Pt must not have neurovascular (nerve/blood vessel) compromise
* Pt must not have an open fracture or visible limb deformity
* Pt must not be a pediatric patient who presents with a gait abnormality of unknown origin.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to an urban and suburban community hospital with acute foot or ankle injury
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
amount of radiographs obtained in the ED. | Participants will be followed for the duration of their ED stay, expected not to be greater than an average of 4 hours
  This study aims to determine if triage application of the OAR and OFR can decrease the amount of radiographs obtained in the ED.

SECONDARY OUTCOMES:
waiting times/length of stay (LOS) | Participants will be followed for the duration of their ED stay, expected not to be greater than an average of 4 hours
  The implementation of the OAR and OFR at triage by the nursing staff is expected to decrease the amount of radiographs obtained in the ED and decrease LOS.

OTHER OUTCOMES:
patient satisfaction with their care in the ED. patient satisfaction with their care in the ED. | Participants will be assessed at the end of their ED stay, expected not to be greater than an average of 4 hours
  It is anticipated that Both patient and provider satisfaction will increase as a result of OAR/OFR implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Marna R Greenberg, DO, MPH, Principal Investigator — Lehigh Valley Hospital
Locations (1):
- Lehigh Valley Hospital and Health Network, Allentown, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD, just publish the study results.